CLINICAL TRIAL: NCT03724188
Title: Impact of Parathyroidectomy on Vascular Calcification and Clinical Outcome in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Mansoura General Hospital (Other)
Responsible Party: Principal Investigator, Nadia Mohsen Abdu Ibrahim, consultant of nephrology, Mansoura General Hospital
Other Study IDs: MD/17.11.133
Record Dates: First submitted 2018-10-24; First posted 2018-10-30 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Hyperparathyroidism, Secondary
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- parathyroidectomy group: the parathyroidectomy group includes 40 hemodialysis patients suffering from sever secondary hyperparathyroidism undergoing surgical parathyroidectomy
  Interventions: Procedure: surgical parathyroidectomy
- non parathyroidectomy group: 15 hemodialysis patients with sever secondary hyperparathyroidism who were indicated for surgical parathyroidectomy but did not underwent surgery and continued on medical treatment

INTERVENTIONS:
Procedure: surgical parathyroidectomy — total parathyroidectomy, subtotal parathyroidectomy, total parathyroidectomy with autotransplantation
  Groups: parathyroidectomy group

SUMMARY:
The aim of this study is to assess the clinical, laboratory and vascular calcification outcome within 6 months duration in patients undergoing surgical parathyroidectomy (total, subtotal, and total with autotransplantation)

DETAILED DESCRIPTION:
All patients above the age of 18, with end stage renal disease maintained on regular hemodialysis and are indicated for surgical parathyroidectomy.

The indications for parathyroidectomy included persistently elevated intact parathormone hormone levels of greater than 500 pg/mL, uncontrolled hypercalcaemia with hyperphosphataemia or clinical symptoms of secondary hyperparathyroidism refractory to medical treatment. These symptoms included bone pain, pruritus, fracture, fatigue and calciphylaxis

These patients will be exposed to pre-operative evaluation of clinical, laboratory and vascular calcification in abdominal aorta and coronary calcium scoring using ECG- gated non contrast CT in hemodialysis patients undergoing parathyroidectomy

Post-operative evaluation of clinical, laboratory and vascular calcification in abdominal aorta and coronary calcium scoring using non contrast CT will be done 6 months post-operative

Assessment of the relation between preoperative and postoperative measures

Patients with the following criteria will be excluded:

1. chronic kidney disease patients not yet on regular Hemodialysis
2. patients who had primary hyperparathyroidism
3. patients who had received kidney transplantation
4. patients who underwent repeated parathyroidectomy
5. patients who were lost to follow-up or with missing data.

ELIGIBILITY:
Inclusion Criteria:

* All patients above the age of 18
* patients with End stage renal disease maintained on regular hemodialysis
* indicated for surgical parathyroidectomy

Exclusion Criteria:

* Chronic kidney disease patients not yet on regular Hemodialysis
* patients who had primary hyperparathyroidism
* patients who had received kidney transplantation
* patients who underwent repeated parathyroidectomy
* patients who were lost to follow-up or with missing data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All patients above the age of 18, with ESRD maintained on regular hemodialysis and are indicated for surgical parathyroidectomy
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
emergent adverse postoperative events and assessment of the degree of vascular calcification | 6 months
  assessment of emergent adverse postoperative events as bleeding, indication for mechanical ventilation and intensive care unit admission, vocal cord injury and development of hypoparathyroidism with persistent hypocalcemia assessment of degree of vascular calcification via measuring calcium scoring through ECG gated non contrast CT

SECONDARY OUTCOMES:
Emergent Adverse events on laboratory parameters | 6 months
  assessment of s.calcium in mg/dl s.phosphorus ( mg/dl) and level of intact parathormone hormone in ( pg/mL)
Emergent Adverse events on Quality of life through assessing physical functioning, limitations due to physical health, limitations due to emotional problems, Energy/Fatigue, Emotional wellbeing, Social functioning, Pain, and General health | 6 months
  Emergent Adverse events on Quality of life using short form 36 heath survey questionaire to assess physical functioning, limitations due to physical health, limitations due to emotional problems, Energy/Fatigue, Emotional wellbeing, Social functioning, Pain, General health
Emergent Adverse events on clinical status of the patient | 6 months
  improvement of clinical symptoms related to hyperparathyroidism prior to surgery, occurrence of surgical complications related to parathyroidectomy procedure, cardiovascular problems, bone aches and disabilities, pruritis

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M Abbas, PhD, Study Chair — Institutional Research Board MFM; Ahmed M Halawa, PhD, Study Chair — Institutional Research Board MFM; . Donia M Sobh, Study Director — Institutional Research Board MFM; Nagy S Abd-elhady, PhD, Study Chair — Institutional Research Board MFM
Locations (1):
- Faculty of medicine - Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
data collection is not yet complete, study is still ongoing for upgrading and expansion